CLINICAL TRIAL: NCT06289426
Title: The Effectiveness of a Yoga Intervention in Improving the Wellbeing and Productivity of Desk-based Workers
Brief Title: Online Yoga for Improving the Well-being of Desk-based Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kingston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KU3339
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Perceived Stress; Depression; Anxiety; Mindfulness; Self-Compassion; Compassion; Work Engagement; Productivity; Heart Rate Variability; Mental Wellbeing; Musculoskeletal Pain
MeSH Terms: conditions — Depression; Anxiety Disorders; Musculoskeletal Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga - Group S (Experimental): The experimental group will participate in 8 weeks of live online yoga classes, 3 times a week for 60 minutes each session. The yoga program will be designed based on previous evidence and personal experience of yoga experts and researchers.
  Interventions: Other: Yoga
- Control - Group L (No Intervention): The control group will be waitlisted and will continue with the usual routine for 8 weeks. They will participate in 8-week yoga classes after the completion of the study.

INTERVENTIONS:
Other: Yoga — The yoga program will consist of body awareness, meditation, poses, breathing practices, relaxation, and positive affirmations in Sanskrit and English.
  Arms: Yoga - Group S

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of an 8-week online yoga intervention in improving the well-being and productivity of desk-based workers. The main questions it aims to answer are:

* How effective is an 8-week online yoga intervention in improving the well-being (mental and physical) and productivity (work engagement and job performance) of the yoga group compared with passive controls?
* Are there any differences in well-being and work-related measures between the yoga and control groups?

Participants in the yoga group will practice yoga three days a week for 8 weeks and will be compared with a wait-listed control group, which will continue with the usual routine for 8 weeks. Researchers will evaluate the impact of yoga on the well-being and productivity of desk-based workers.

DETAILED DESCRIPTION:
Office workers are reported to spend 75% of their working day sitting (Mansoubi et al., 2016) and up to 10 hours across the whole day on workdays (Clemes et al., 2014). This presents a significant challenge to workforce well-being because of the increasing prevalence of remote work globally. A recent survey by the Office for National Statistics found that as of November 2022, the top four sectors in the UK using, or intending to use, increased homeworking as a permanent business model were those consisting of desk-based or office workers as their employees; viz information and communication (43.3%), professional scientific and technical activities (29.4%), education (17.2%), and administrative and support service activities (14.3%) (Office for National Statistics (ONS), 2022).

The most common problems among desk-based workers compared to any other occupational groups include the musculoskeletal symptoms of the neck and shoulders, wrists and hands, lower back, and upper extremities (AlOmar et al., 2021; Basakci Calik et al., 2022; Besharati et al., 2020; Bontrup et al., 2019; Mohammadipour et al., 2018). Furthermore, high sedentary behaviour is also associated with a greater risk of anxiety (Teychenne et al., 2015), depression (Hallgren et al.; Wang et al., 2019), perceived stress, particularly in white-collar employees (Dėdelė et al., 2019), adverse mental health (Hamer et al., 2014), lower job satisfaction and greater fatigue (Rosenkranz et al., 2020). Office workers, in particular, have been found to have a higher prevalence of common mental health disorders compared to other occupations in the UK (Stansfeld et al., 2011). Work-related ill health is also a significant concern for employers because of the productivity loss resulting in a substantial financial burden to the organizations (Griffiths et al., 2011; Johnston et al., 2008).

Yoga has been accepted as a holistic practice similar to mindfulness with the added advantage of components like postures (asana) and breathing practices (pranayama), providing physical, mental, emotional, social, and spiritual benefits (Gordon, 2013; Vergeer et al., 2021). As a multi-component practice, yoga can provide a holistic approach to managing the consequences of prolonged desk-based work. It appears to be a suitable and safe therapy that may improve pain and functional outcomes connected to a range of musculoskeletal conditions in a clinically relevant manner (Ward et al., 2013). Yoga has also shown positive effects on the mental health of various employee types, including office workers, as per two systematic reviews and a meta-analysis (Valencia et al., 2019; Valle et al., 2020). The rising prevalence of desk-based work and its likelihood of representing a larger proportion of the future workforce underlines the timeliness of this study.

Therefore, the study aims to explore the effectiveness of an 8-week yoga intervention in improving the well-being (mental and physical) and productivity (work engagement and job performance) of the yoga group compared with passive controls.

ELIGIBILITY:
Inclusion Criteria:

1. Participants working remotely/hybrid aged 18 years and above.
2. living and working in the UK.
3. speak and understand English.
4. Fulfil the health criteria (e.g., No current injuries ).
5. Are willing to commit to an 8-week online streamed yoga course, three times a week, 60 min each session

Exclusion Criteria:

1. Current yoga practice or related activities.
2. Medical or psychiatric conditions limiting the practice of yoga in general
3. Not suffering from any serious medical or psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | 8 Weeks
  The questions in this scale ask about your feelings and thoughts during the last month. In each case, you will be asked to indicate how often you felt or thought a certain way.
PROMIS-Anxiety Short form | 8 Weeks
  The 7-item PROMIS Anxiety Short Form assesses the pure domain of anxiety in individuals age 18 and older.
The Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) | 8 Weeks
  The SWEMWBS is a short version of the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS). The WEMWBS was developed to enable the monitoring of mental wellbeing in the general population and the evaluation of projects, programmes and policies which aim to improve mental wellbeing.
The Mindful Attention Awareness Scale (MAAS) | 8 Weeks
  The trait MAAS is a 15-item scale designed to assess a core characteristic of mindfulness, namely, a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present, simply observes what is taking place.
The Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) | 8 Weeks
  The Cornell questionnaire was used to determine the level of pain among office employees in response to rest breaks and ergonomic modifications. Musculoskeletal discomforts, particularly pain severity among office employees, can be collected by the Cornell questionnaire shown to be a valid and reliable tool.
Self-Compassion Scale Short Form (SCS-SF) | 8 Weeks
  The Self-Compassion Scale - Short Form (SCS-SF) is a 12-item self-report measure that is used by adults to measure their capacity for self-compassion - the ability to hold one's feelings of suffering with a sense of warmth, connection and concern.
The Compassion Scale (CS) | 8 Weeks
  The CS has the same general structure as the SCS and measures compassion for others.
Uterecht Work Engagment Scale-Short Form (UWES -9) | 8 Weeks
  The UWES utilizes three scales to determine the level of work engagement:
  Vigor, dedication, and absorption. It is a test of how to measure work engagement both on an individual and on group level: vigor, dedication, and absorption.
Work Ability Index (WAI) | 8 Weeks
  It measures current work ability compared to highest work ability ever.
Center for Epidemiologic Studies Short Depression Scale (CES-D-R 10) | 8 Weeks
  This scale is a self-report measure of depression.
Heart Rate Variability (HRV) | 8 Weeks
  HRV is simply a measure of the variation in time between each heartbeat. This variation is controlled by a primitive part of the nervous system called the autonomic nervous system (ANS). It works behind the scenes, automatically regulating our heart rate, blood pressure, breathing, and digestion among other key tasks. But in recent years, companies have launched apps and wearable heart rate monitors that monitor HRV. We are using a Polar H10 heart rate sensor to measure HRV of participants to see physiological changes in stress levels due to practising yoga.

CONTACTS AND LOCATIONS:
Overall Officials: Vipin Wadhen, MPhil, Principal Investigator — Kingston University
Locations (1):
- Vipin Wadhen, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July 2025
Access Criteria: Individual Participant Data (IPD) will be available upon reasonable request to qualified researchers. Data-sharing requests must be submitted in writing to the principal investigator and will be evaluated based on the scientific merit and ethical considerations of the proposed analysis. Access will be granted for purposes related to the exploration of well-being, productivity, or similar fields in desk workers or yoga interventions. Approved researchers must sign a data-sharing agreement and ensure the confidentiality and appropriate use of the data. Data will be provided through a secure repository, and access will be granted for a limited period. Requests will be reviewed by a data access committee, which will assess proposals based on their relevance to the research area and potential contribution to the field.